CLINICAL TRIAL: NCT06806085
Title: Analysis of Influencing Factors of High-Order Aberrations of Small Incision Lenticule Extraction with Lenticule Retained
Brief Title: Analysis of Influencing Factors of High-Order Aberrations of SMILE with Lenticule Retained
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Jian Xiong, Associate research fellow; Attending physician, Second Affiliated Hospital of Nanchang University
Other Study IDs: [2024] NO.(138)
Record Dates: First submitted 2025-01-26; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-10

CONDITIONS: Small-incision Lenticule Extraction (SMILE) Surgery; Corneal Higher-order Wavefront Aberrations; Residual Lenticule
Keywords: Residual Lenticule; Corneal Higher-order Wavefront Aberrations; Small-incision Lenticule Extraction
MeSH Terms: conditions — Smiling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- lenticule retained group
- Non-lenticule retained group

SUMMARY:
Analysis of Influencing Factors of High-Order Aberrations of SMILE with Lenticule Retained

DETAILED DESCRIPTION:
Wavefront analysis and other objective methods are the mainstream approaches for assessing visual quality after refractive surgery, with high-order aberrations being the main observation indicators. Some studies have explored the correlation between various complications after SMILE surgery and high-order aberrations. However, research on lenticule retained after surgery has mainly focused on clinical management and case reports of overt lenticule retained, while there is a lack of high-quality observational studies on the population with covert lenticule retained (periphery residual lenticule) to serve as evidence. This often puts clinicians in a dilemma of whether to perform another surgery to remove the remnants. In summary, although research on lenticule retained after SMILE surgery is gradually increasing, systematic studies on their relationship with higher-order aberrations are still insufficient. This study aims to fill the gap in existing research by comparing and analyzing high-order aberrations between patients with and without periphery residual lenticule, providing a more comprehensive assessment of postoperative visual quality. This will offer important theoretical basis and practical guidance for improving SMILE surgical techniques and optimizing postoperative management.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, gender unrestricted;
2. Equivalent spherical refraction ≤ -10.0D, corrected distance visual acuity ≥ 1.0, myopia stable for ≥ 2 years, and no contact lens wear for at least 2 weeks;
3. The patient voluntarily participates in this study, signs the informed consent form, and agrees to follow up according to the study plan;
4. Predicted postoperative residual corneal stromal thickness ≥ 280 micrometers.

Exclusion Criteria:

1. Subclinical keratoconus, keratoconus, moderate to severe corneal opacities or scars, and other ocular conditions;
2. Diabetes, keloid-prone constitution, autoimmune and connective tissue diseases, etc.;
3. Severe mental disorders such as generalized anxiety disorder, panic disorder, depression, schizophrenia, and bipolar disorder; inability to cooperate with physicians;
4. Refusal to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Each subject must have complete surgical video recordings and medical records.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Δ Higher-order Aberration | Day 90
  Preoperative and postoperative Higher-order aberration difference obtained from wavefront aberrations map of corneal topography in Pentacam measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No